CLINICAL TRIAL: NCT04158024
Title: The Effect of Erector Spinae Plane Block on Neurodevelopmental Outcomes of Neonatal Congenital Heart Disease Patients
Brief Title: Erector Spinae Plane Block in Congenital Heart Disease Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 53993
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Congenital Heart Disease in Children; Neurologic Complication
Keywords: Erector Spinae Plane Blockade; Pediatric Congenital Heart Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volatile Anesthetic Control (No Intervention): In volatile anesthetic technique, maintenance of anesthesia will be standardized to the volatile anesthetic isoflurane. Isoflurane will be delivered at 1.5-2.0%% as required for anesthetic management.
  Rocuronium or pancuronium will be used for muscle relaxation. Narcotic, fentanyl will be administered at no greater than 2 mcg/kg/hr. However, the primary anesthetic during CPB will be isoflurane with no narcotic administered during CPB.
- Erector Spinae Plane Blockade Treatment (Experimental): Patients will receive an erector spinae plane blockade prior to their surgery as per standard regional anesthesia technique in addition to the standard of care Volatile Anesthetic Treatment.
  Interventions: Other: Erector Spinae Plane Block

INTERVENTIONS:
Other: Erector Spinae Plane Block — The ESPB is a fascial plane block performed by injecting local anesthetic between the erector spinae muscle and the transverse process. Its proposed mechanism of action is via blockade of the dorsal and ventral rami of the thoracic spinal nerves and sympathetic fibers.
  Arms: Erector Spinae Plane Blockade Treatment

SUMMARY:
Pediatric cardiac patients undergoing surgical anesthesia are at an increased risk of poor neurologic outcome (20-50%). Unattenuated anesthetic exposure and pain contributes to physiologic perturbations that may increase neurologic morbidity. Because of the often-large exposure to anesthetic agents in these cardiac children, at such a young age and the potential modifying anesthetic practice that could lead to improved neurodevelopmental outcomes and surgical recovery is paramount. Regional anesthesia such as thoracic epidurals provide effective analgesia and reduced intraoperative anesthetic needed but carry devastating sequelae neurological risks of epidural hematomas after anticoagulation during cardiopulmonary bypass (CPB). Recently, a newly described erector spinae plane block (ESPB) is superficial to neuraxial or vascular structures, providing opportunity to be placed with less risk for surgery requiring CPB. This block has been described as effective regional anesthesia for adult cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Neonates of at least 32 weeks of gestation, infants and children admitted to The Lucile Packard Children's Hospital for treatment of cyanotic or non-cyanotic heart disease requiring surgical intervention.
* Admitting diagnosis of cyanotic or non-cyanotic heart disease

Exclusion Criteria:

* Neonates less than 32 weeks of gestational age
* Any documented central nervous system malformations.
* Any potential subject requiring unexpected postoperative Extracorporeal membrane oxygenation (ECMO) support

Ages: 32 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Length of Stay (LOS) | Through hospital stay, an average of 5 days
  Determine if bilateral surgical placed ESPBs will decrease length of stay in the pediatric ICU and the hospital. LOS and decrease postoperative opioid consumption.)
Postoperative Opioid Consumption | Through hospital stay, an average of 5 days
  Determine if bilateral surgical placed ESPBs will decrease postoperative opioid consumption measured in Morphine Milligram Equivalents (MME)
Comparing Changes in EEG Monitoring | Pre-operatively and up to 48 hours prior to discharge
  Evaluate the changes in EEG waves from measurements performed prior to induction of anesthesia to those collected following the procedure to definitively determine abnormalities in the EEG. The EEG will monitor the Alpha, Beta, Delta, and Theta bandwidths to determine an abnormality.
Neurological and Neurobehavioral Testing - Bayley III | 12-48 Months Post-Operatively
  Evaluate long-term neurological outcomes as per standard of care testing including the Bayley Exam III
Neurological and Neurobehavioral Testing - Capute Scale | 12-48 Months Post-Operatively
  Evaluate long-term neurological outcomes as per standard of care testing including the and Capute Scales. Scores 86 and higher represent typical neurological development. Scores between 71 and 85 represent borderline delays. Scores 70 or lower indicate significant delays in development.

SECONDARY OUTCOMES:
Choline | 0-72 Hours
  Blood Levels
Glutamate | 0-72 Hours
  Blood Levels
N-Acetylaspartate | 0-72 Hours
  Blood Levels
Lactate | 0-72 Hours
  Blood Levels

IPD SHARING:
Plan to Share IPD: No